CLINICAL TRIAL: NCT04304404
Title: The Effect of Risk Reduction Program Applied to Women With High Breast Cancer Risk on Participation in Screening, Health Beliefs and Behavior
Brief Title: Risk Reduction Program for Women Having High Risk of Breast Cancer
Acronym: BrCaRRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Habibe ÖZÇELİK, Lecturer, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 68824072019
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Cancer Screening; Early Detection of Cancer; Breast Cancer; Preventive Health Care; Health Behavior
MeSH Terms: conditions — Breast Neoplasms; Health Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (BrCaRRP) (Experimental): Individual interventions based on the Health Belief Model and the The Health Promotion Model involving education, guidance, counseling, case management and surveillance for women with high breast cancer risk
  Interventions: Behavioral: Breast Cancer Risk Reduction Program (BrCaRRP)
- Control Group (No Intervention): An information note will be given to the control group. The post-tests will be collected at the end of 12 weeks

INTERVENTIONS:
Behavioral: Breast Cancer Risk Reduction Program (BrCaRRP) — Women in the intervention group will complete the pre-tests electronically, and a 12-week intervention program will be implemented. The first meeting will be face-to-face individual training. In this training session, the risk of developing breast cancer will be calculated with each participant using breast cancer risk assessment tools. Modifiable and non-modifiable factors that increase breast cancer risk will be explained. With the participant, it will be decided which of the modifiable risk factors will be improved. Guidance will be given on topics such as genetic counseling, breast cancer screenings, increasing physical activity, healthy nutrition, weight control, smoking and alcohol use. The interventions will continue with phone calls and the 12-week program will be completed.
  Other Names: İntervention Group (BrCaRRP)
  Arms: Intervention group (BrCaRRP)

SUMMARY:
An intervention program involving education, guidance, counseling, case management and surveillance based on the Health Belief Model will be implemented on women with high risk of breast cancer. The impact of the breast cancer risk reduction program on participation in breast cancer screenings, health beliefs (health motivation, sensitivity, fear of breast cancer) and behaviors (physical activity, nutrition, health responsibility, genetic counseling) will be evaluated in the study.

DETAILED DESCRIPTION:
In women with family history of breast cancer, cancer risk increases at least twice as compared to the population of the same age. The aim of this study is to evaluate the impact of the intervention program based on the Health Belief Model involving education, guidance, counseling, case management and surveillance, on participation in breast cancer screenings, health beliefs and behaviors in women with high risk of breast cancer.

This study protocol describes a randomized controlled trial with parallel group design. First degree biological relatives (mother, daughter, sister) of breast cancer patients who are diagnosed with breast cancer at or under the age of 50 and who apply to the Oncology Department will be randomly assigned to the intervention and control group.

The content of the Breast Cancer Risk Reduction Program created for the Intervention Group was planned according to the Health Belief Model (HBM) theoretical framework. The interventions based on HBM were carried out according to the OMAHA nursing interventions categories used in the field of Public Health Nursing (training, guidance, counseling, case management and surveillance). Breast Cancer Risk Reduction Program (BirCarrePro) is a 12-week program that includes six interviews. The first intervention in this group will begin with a 60-minute face-to-face individual training. After the first face-to-face interview, phone calls will be made in the second, third, sixth, ninth, and twelfth weeks. Pre-tests and post-tests will be completed by the participants via electronic questionnaires. Follow-up questionnaires will be applied by repeating the post-test at the 24th week. In the control group, post-test will be applied 12 weeks after the pre-test, and follow-up questionnaires will be applied 24 weeks after the pre-test.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being the first degree biological relative of a primary breast cancer patient diagnosed at or before the age of 50
* Aged 25 or older
* No mammography and/or MRI in the last 18 months
* Being literate

Exclusion Criteria:

* Having been diagnosed with breast cancer (first degree relative)
* Being pregnant or breastfeeding

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Breast Cancer Screening | 12 weeks
  The primary outcome measure of the study is the participation rate of first degree relatives in breast cancer screenings.
Health Belief Model Scale (Susceptibility, Health Motivation sub-factors) | 12 weeks
  Health Belief Model Scale (Susceptibility, Health Motivation sub-factors)Health Motivation' sub-dimensions of Champion's Health Belief Model Scale will be used in this study. Sensitivity sub-dimension consists of 3 items, and Health Motivation sub-dimension consists of 5 items. In this 5-point Likert type scale, the items are scored as follows: "totally disagree" (1), "disagree" (2), "undecided" (3), "agree" (4), "totally agree" ( 5). All items of this scale are positive. Total score ranges from 8 to 40. Higher scores indicate higher sensitivity and health motivation. The scale contains no reverse items.
Breast Cancer Fear Scale | 12 weeks
  Champion's Breast Cancer Fear Scale consists of two sub-dimensions and eight items. It consists of five items related to thought and three items related to physiological stimulation. In this 5-point Likert type scale, the items are scored as follows: "totally disagree" (1), "disagree" (2), "undecided" (3), "agree" (4), "totally agree" (5). Total score ranges from 8 to 40. As the score increases, the level of breast cancer fear increases. The scale contains no reverse items.
Healthy Lifestyle Behaviors Scale II (Health Responsibility, Physical Activity and Nutrition Sub-Scale) | 12 weeks
  All items of the Healthy Lifestyle Behaviors Scale are positive and are structured as 4-point Likert type items. The scoring is as follows: never (1), sometimes (2), often (3), regularly (4). The scale consists of six sub-dimensions. Only 'Health Responsibility, Physical Activity and Nutrition' sub-dimensions were used in this study. The lowest score that can be obtained from these three sub-dimensions is 26 and the highest score that can be obtained is 104. Higher scores indicate more healthy lifestyle behaviors.
International Physical Activity Questionnaire (IPAQ) | 12 weeks
  IPAQ short form that will be used in this study consists of four sub-dimensions (Severe Physical Activity, Moderate Physical Activity, Mild Physical Activity, and Sitting Times) and seven items. The time spent on mild, moderate and severe activities as well as sitting times and the energy spent in these activities are calculated. The severity, frequency and duration of the activities performed for 10 minutes or longer in the last seven days are evaluated and the activity level is determined as metabolic equivalent (MET). Walking is 3.3 MET, moderate to severe physical activity is 4.0 MET, and severe physical activity is 8.0 MET. The 'MET-min/week' value is obtained by multiplying the MET value of each physical activity level with the days and minutes this physical activity is performed every week. The obtained MET value is classified as severe physical activity (MET>3000), moderate physical activity (MET = 600-3000), and mild physical activity (MET <600).

CONTACTS AND LOCATIONS:
Overall Officials: Sebahat GÖZÜM, Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ozcelik H, Gozum S. The Effect of the Breast Cancer Risk Reduction Program on Women With High Breast Cancer Risk in Terms of Their Participation in Screening and Their Health Beliefs and Behavior: A Study Protocol for a Randomized Controlled Trial. Cancer Nurs. 2024 Nov-Dec 01;47(6):E376-E386. doi: 10.1097/NCC.0000000000001229. Epub 2023 Mar 13. PMID 36907899